CLINICAL TRIAL: NCT02756351
Title: A Double-blinded Randomized Clinical Pilot Trial of Nasal Prongs With Proprietary Surface Coating Aiming to Reduce Bacterial Colonization
Brief Title: A Efficacy and Safety Study of Nasal Prongs With Proprietary Surface Coating Aiming to Reduce Bacterial Colonization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CytaCoat AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CCNP-01
Record Dates: First submitted 2016-04-26; First posted 2016-04-29 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Nosocomial Infections; Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Cross Infection; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- CytaCoat Nasal Prong (Experimental): The CytaCoat Nasal Prong is composed of the reference device coated with CytaCoat technology.
  Interventions: Device: CytaCoat Nasal Prong
- Reference Nasal Prong (Active Comparator): Inspiration Healthcare Inspire nCPAP Nasal Prong consists of silicone. Is a Conformité Européenne marked (CE-marked) commercially available medical device.
  Interventions: Device: Inspiration Healthcare Inspire nCPAP Nasal Prong

INTERVENTIONS:
Device: CytaCoat Nasal Prong
  Arms: CytaCoat Nasal Prong
Device: Inspiration Healthcare Inspire nCPAP Nasal Prong
  Arms: Reference Nasal Prong

SUMMARY:
The study is a first step in establishing the safety and efficacy of the CytaCoat technology when applied to a medical device such as a nasal prong and the clinical data generated will serve as a basis for continuous studies in clinically significant settings such as the neonatal care units.

ELIGIBILITY:
Inclusion Criteria:

1. Legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the informed consent form (ICF).
2. Subject is between 18 and 65 years of age.
3. Subjects that have intact, wound free and scar free skin at the Nasal Prong target site.
4. Subject that have intact, irritation-free nasal mucus membrane.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Subjects who are active smokers or using snuff.
3. Subjects currently suffering from a common cold, sinusitis, allergies or sleep apnea.
4. Subjects suffering from and/or subjects that have experienced nosebleed within 1 month prior to entering the study.
5. Subjects using and/or subjects that have used oral or topical antibiotics within 2 weeks prior to entering the study.
6. Subjects using and/or subjects that have used oral or topical anti-inflammatory drugs within 1 week prior to entering the study.
7. Subjects participating in any other clinical study.
8. Subjects diagnosed with any type of skin infection (bacterial, viral or fungal) or inflammatory skin disease including psoriasis, eczema or severe acne
9. Subjects diagnosed with any type disease affecting mucus membranes.
10. Subjects suffering from any other condition or symptoms preventing the subject from entering the study, according to the investigator´s judgment.
11. Subjects who have a lesion (including lymphadenopathy), dysaesthesia, previous surgery or abnormal anatomy at the Nasal Prong target site
12. Any subject that according to the Declaration of Helsinki is deemed unsuitable for study enrolment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baldvin Jonsson, Principal Investigator — Neonatal, Karolinska University Hospital
Locations (1):
- Neonatal, Karolinska University Hospital, Stockholm, Stockholm County, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- CytaCoat Nasal Prong: The CytaCoat Nasal Prong is composed of the reference device coated with CytaCoat technology.
  CytaCoat Nasal Prong
- Reference Nasal Prong: Inspiration Healthcare Inspire nCPAP Nasal Prong consists of silicone. Is a Conformité Européenne marked (CE-marked) commercially available medical device.
  Inspiration Healthcare Inspire nCPAP Nasal Prong
Period: Overall Study
Arm/Group | CytaCoat Nasal Prong | Reference Nasal Prong
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CytaCoat Nasal Prong | Reference Nasal Prong | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.96 (14.22) | 31.58 (13.44) | 32.77 (13.74)
Gender [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  Sweden | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Bacterial Colonization of the Nasal Prong After 18 Hours of Device Usage When Comparing the CytaCoat Nasal Prong to the Reference Device.
Time Frame: 18 hours
Measure: Mean (Standard Deviation); unit: fold change in log value
Arm/Group | CytaCoat Nasal Prong | Reference Nasal Prong
Number analyzed (Participants) | 24 | 24
fold change in log value | 8.29 (4.40) | 21.69 (1.93)

2. Secondary Outcome: Any Adverse Events Such as Skin Reactions, Allergic Reactions, Abrasions, Shears or Wounds Due to Contact or Pressure of the Device on the Nose of Subjects Occurring During the Study.
Time Frame: 18 hours
Measure: Number; unit: Adverse Events
Arm/Group | CytaCoat Nasal Prong | Reference Nasal Prong
Number analyzed (Participants) | 24 | 24
Adverse Events | 24 | 23

ADVERSE EVENTS:
Time Frame: Adverse Events were reported throughout the study, i.e. 15 March until 28 June 2016. For each subject Adverse Events were reported until the subject had completed the study, e.g. between Visit 1 and 2 (18 hours of participation). One subject was followed- up one extra day before the Adverse Event was assessed as resolved.
Arm/Group | CytaCoat Nasal Prong | Reference Nasal Prong
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 17/24 | 16/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CytaCoat Nasal Prong (N=24) | Reference Nasal Prong (N=24)
Mark on columella (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5)
Pain (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Mark on tip of the nose (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Itch (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Breathing problems (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Breathing problems due to extra Steri-Strips put over the device.
Humidity (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Irritation and sore (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Itch and humidity (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Mark (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Psychological (Social circumstances) | 1 (1) | 1 (1)
Sore (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Stingy (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Breathing problems and itch (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Irritation and stingy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sleepwalking, nausea and a feeling of fainting (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As stated in the Clinical Investigation Plan (CIP):

The Principal Investigator may publish results from this investigation; however as some of the information regarding the investigational medical device and development activities may be of a strictly confidential nature, the Sponsor must first be given the opportunity to review any publication manuscript prior to submission to journals, meetings or conferences.